CLINICAL TRIAL: NCT06011460
Title: Observation of Clozapine Treatment Safety in Bipolar Disorder.
Acronym: CloGD
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: NKBBN/355-183/2023
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Bipolar Disorder
Keywords: clozapine; bipolar disorder; suicidality; adverse events
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation | interventions — Clozapine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients' name: Diagnosis of treatment-resistant depressive episode in the course of bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders-5. Age from 18 to 65 years old.
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Clozapine — Diagnosis of treatment-resistant depressive episode in the course of bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
  Age from 18 to 65 years old.

SUMMARY:
The purpose of the registry is to record incidence of adverse events during treatment with clozapine in patients suffering from bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder, with its spectrum, remains a life-long and significant mental health concern due to its unpredictable nature and varied symptomatology. Despite the wide array of available treatments, some cases of bipolar disorder remain resistant to traditional medications. Clozapine, traditionally used for treatment-resistant schizophrenia, has shown promising results in managing resistant cases of bipolar disorder, particularly reducing the risk of suicide. There are not enough controlled studies on clozapine, especially in treatment resistant bipolar depression.

There are certain limitations associated with the use of clozapine, primarily related to the possibility of adverse events including agranulocytosis, myocarditis, pneumonia, intestinal obstruction and seizures. Therefore, there is a need for more studies on safety and tolerability of this treatment in patients with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of treatment-resistant depressive episode in the course of bipolar disorder according to DSM-5.
* Age from 18 to 65 years old.

Exclusion Criteria:

* Patients unable to give fully written informed consent
* Patients unable to comply with the requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bipolar disorder treated with clozapine.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety measures of clozapine treatment in patients with bipolar disorder. | 1 year
  Incidence of possible occurrence of adverse events during treatment with clozapine in patients with bipolar disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Wiesław J Cubała, M.D. PhD, Principal Investigator — Medican University of Gdańsk
Locations (1):
- Department of Psychiatry, Medical University of Gdańsk, Gdansk, Pomeranian Voivodeship, Poland

REFERENCES:
- [Background] Wilkowska A, Wiglusz MS, Cubala WJ. Clozapine: promising treatment for suicidality in bipolar disorder. Psychiatr Danub. 2019 Sep;31(Suppl 3):574-578. PMID 31488793
- [Background] Wilkowska A, Cubala WJ. Clozapine As Transformative Treatment In Bipolar Patients. Neuropsychiatr Dis Treat. 2019 Oct 9;15:2901-2905. doi: 10.2147/NDT.S227196. eCollection 2019. PMID 31632038
- [Background] Wilkowska A, Wiglusz MS, Cubala WJ. Clozapine in Treatment-Resistant Bipolar Disorder With Suicidality. Three Case Reports. Front Psychiatry. 2019 Jul 19;10:520. doi: 10.3389/fpsyt.2019.00520. eCollection 2019. PMID 31379632
- [Background] Delgado A, Velosa J, Zhang J, Dursun SM, Kapczinski F, de Azevedo Cardoso T. Clozapine in bipolar disorder: A systematic review and meta-analysis. J Psychiatr Res. 2020 Jun;125:21-27. doi: 10.1016/j.jpsychires.2020.02.026. Epub 2020 Feb 27. PMID 32182485